CLINICAL TRIAL: NCT03382275
Title: EXPLorative Data Collection for Patient chAracterIzation, treatmeNt Pathways and Outcomes of IRON Preparations
Acronym: EXPLAIN-IRON
Status: Completed | Type: Observational
Sponsor: GWT-TUD GmbH (Other)
Collaborators: Shield Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: EXPLAIN IRON
Record Dates: First submitted 2017-12-12; First posted 2017-12-22 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Iron-Dextran Complex; ferric maltol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Iron Supplement — any oral or intravenous prescription iron supplement
  Other Names: Iron bivalent or trivalent oral; Iron trivalent oral; Feraccru (Ferric Maltol)

SUMMARY:
By describing the characteristics of iron deficiency (ID) patients treated with various oral or intravenous iron formulations and their outcomes, this registry will provide the medical community with important information to support treatment decisions for their patients regarding data on effectiveness, safety, tolerability, treatment persistence, quality of life, and therapeutic costs. This will ultimately support improvements to patient care, including the long-term outcomes of patients with ID.

DETAILED DESCRIPTION:
Iron deficiency (ID) anaemia is a prevalent condition in Germany and other Western countries. It is a common complication in inflammatory bowel disease (IBD), cardiovascular disease including chronic heart failure, cancer, chronic kidney disease (CKD), gynaecological conditions, and others.

Anaemia has a strong impact on patient's quality of life and ability to work, and removing the condition by increasing the haemoglobin may improve QoL and other patient-related outcomes. While in certain patient groups, such as CKD, anaemia is addressed on a routine basis, in others it remains widely undertreated. For example, in IBD patients across various European countries, iron supplementation was administered in only up to 28% of individuals.

For iron supplementation aimed to replenish to body' iron stores, there are numerous oral, and intravenous preparations available.

The most convenient approach is oral administration, where Fe2+ salts are mostly used. Usually low doses between 50 - 100 mg daily are recommended, as the duodenum can only absorb 10 - 20 mg daily, and higher doses are associated with gastrointestinal side effects including diarrhoea, nausea, flatulence and gastric erosions. To reduce these common side effects, Fe3+ formulations like ferric maltol (Feraccru) have been newly introduced.

Intravenous preparations are all Fe3+ oxyhydroxides with a carbohydrate coat (iron dextran, gluconate, sucrose, carboxymaltose, or ferumexytol). These preparations are typically used second-line in patients with ID who had unsatisfactory treatment results under oral treatment. IV iron infusions have been associated with hypophosphataemia and hypersensitivity reactions. However these events depend on the preparation and are infrequent.

EXPLAIN-IRON has been set up as the first interdisciplinary registry to add further information on the situation and management of patients who receive iron substitution in various indications: IBD, chronic kidney disease, cancer- or therapy-induced ID, gynaecological conditions (hypermenorrhoea, post-partum, fatigue), cardiological indications (congenital heart disease; chronic heart failure) and other causes of ID.

The registry will allow for documentation of all approved oral and IV preparations. As the registry also serves the specific purpose to collect data on the newly introduced preparation Feraccru (oral ferric maltol), about half of the patient population will be treated with that agent.

The registry will be of interest to assess to which extent the various guidelines on iron substitution have been adopted in clinical practice. Overall, EXPLAIN-IRON is expected to provide a comprehensive picture on the use and the outcomes of iron substitution in Germany. By describing the characteristics of ID patients treated with various iron formulations and their outcomes, this registry will provide the medical community with important information to support treatment decisions for their patients regarding data on effectiveness, safety, tolerability, treatment persistence, quality of life, and therapeutic costs. This will ultimately support improvements to patient care, including the long-term outcomes of patients with ID.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients, aged at least 18 years
* Clinical diagnosis of iron deficiency according to treating physician
* Decision to treat with an oral or intravenous iron supplementation made by treating physician considering the indications of the respective Summary of Product Characteristics (prescribing information)
* maintenance or newly initiated treatment (including returning quitters)
* written informed consent

Exclusion Criteria:

* patient not available for long-term documentation
* concomitant or planned participation in a clinical trial (on iron supplementation)
* concomitant over-the-counter iron supplementation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with iron deficiency in one of the following indications:
  (i) Inflammatory bower disease, (ii) chronic kidney disease, (iii) cancer- or therapy-induced iron deficiency, (iv) gynaecological conditions (hypermenorrhea, post-partum, fatigue), (v) cardiology (including iron deficiency in patients with congenital heart disease or chronic heart failure), and (vi) diverse other causes of iron deficiency.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-04-20 (Actual)

PRIMARY OUTCOMES:
Hemoglobin | at 3 months
  serum level change compared to baseline

SECONDARY OUTCOMES:
Ferritin | at 3 months
  serum level change compared to baseline
Hemoglobin | 2 years
  time to normalisation
Ferritin | 2 years
  time to normalisation

OTHER OUTCOMES:
Transferrin saturation | at 3 months
  Time to normalisation
Adverse events | 2 years
  Type, severity and time of adverse events that are related to and caused by iron treatment (in the physician's opinion)
Hypophosphatemia | 2 years
  Percentage of patients
Self-assessed Quality of life | 2 years
  course over time, by Euroquol five-dimensional questionnaire
Fatigue | 2 years
  course over time, by fatigue-specific FACIT questionnaire
Discontinuation of iron supplementation | 2 years
  Rate of patients
Economic parameters | 2 years
  costs for days of hospitalisation and for physician contacts
Patient satisfaction | 2 years
  Patients' Treatment Satisfaction for Medication (TSQM-9 questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: David Pittrow, MD, PhD, Study Director — GWT-TUD GmbH; Stefan Schreiber, MD, PhD, Principal Investigator — Klinik für Innere Medizin I, Universitätsklinikum Kiel
Locations (2):
- Germany (2):
  - Praxis für Gastroenterologie, Berlin
  - Klinik für Innere Medizin I des Universiätsklinikums, Kiel

IPD SHARING:
Plan to Share IPD: No